CLINICAL TRIAL: NCT04667871
Title: Effect of Cataract Hyperemulsification Surgery on Meibomian Gland Morphology and Function
Status: Withdrawn | Type: Observational
Why Stopped: An six-month follow-up was completed after the treatment
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: XZZ-meibomian gland
Record Dates: First submitted 2020-10-04; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Meibomian Gland Dysfunction
Keywords: meibomian gland; cataract surgery
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eyes for cataract surgery: Eyes for cataract surgery
  Interventions: Procedure: cataract surgery
- Eyes without cataract surgery: Eyes without cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — Eyes for cataract surgery
  Groups: Eyes for cataract surgery

SUMMARY:
50 participants at Eye Hospital of Wenzhou Medical University during August, 2017 to July, 2020 will be enrolled in this study. To study the effect of cataract supermammary surgery on the morphology and function of meibomian glands

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with xerophthalmia
* Undergoing cataract hyperemulsification surgery

Exclusion Criteria:

* No history of ocular surgery and trauma
* Any eye diseases except xerophthalmia
* No treated for xerophthalmia before
* Successful completion of follow-ups

Ages: 38 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients who undergoing cataract hyperemulsification surgery and previously untreated with xerophthalmia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
OSDI scale survey | 08/2017 to 07/2020
  OSDI scale survey
tear meniscus height（mm） | 08/2017 to 07/2020
  tear meniscus height（mm）
first tear film rupture time（s） | 08/2017 to 07/2020
  first tear film rupture time（s）
average tear film rupture time（s） | 08/2017 to 07/2020
  average tear film rupture time（s）
the range of meibomian gland missing（%） | 08/2017 to 07/2020
  the range of meibomian gland missing（%）
meibomian gland average diameter (mm) | 08/2017 to 07/2020
  meibomian gland average diameter (mm)
meibomian gland length (mm) | 08/2017 to 07/2020
  meibomian gland length (mm)
meibomian gland area (mm^2) | 08/2017 to 07/2020
  meibomian gland area (mm^2)
meibomian gland deformation coefficient | 08/2017 to 07/2020
  meibomian gland deformation coefficient
meibomian gland total proportion of glands (%) | 08/2017 to 07/2020
  meibomian gland total proportion of glands (%)
meibomian gland imaging value | 08/2017 to 07/2020
  meibomian gland imaging value

IPD SHARING:
Plan to Share IPD: Undecided